CLINICAL TRIAL: NCT03456219
Title: Determination of Protocol of Nocturnal Food Intake of Shift Workers: a Crossover Randomized and Controlled Study.
Brief Title: Determination of Protocol of Nocturnal Food Intake of Shift Workers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Cibele Aparecida Crispim, Principal investigator, Federal University of Uberlandia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CEP UFU 2250027/2017
Record Dates: First submitted 2018-01-26; First posted 2018-03-07 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Shift Work Type Circadian Rhythm Sleep Disorder
Keywords: Food intake; Sleep; Shift work; Postprandial metabolic response
MeSH Terms: interventions — Diet, High-Protein

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shift workers (Experimental): Night workers of the Hospital of Clinics of Uberlândia, Federal University of Uberlândia, received the normal protein diet.
  Interventions: Other: Normal protein diet
- Night workers (Experimental): Night workers of the Hospital of Clinics of Uberlândia, Federal University of Uberlândia, received the high-protein diet.
  Interventions: Other: High-protein diet

INTERVENTIONS:
Other: Normal protein diet — The intervention with the control diet was composed of 65% of carbohydrates, 15% of proteins and 20% of lipids.
  Arms: Shift workers
Other: High-protein diet — The intervention with the higher-protein diet was composed of 45% of carbohydrates, 35% of proteins and 20% of lipids.
  Arms: Night workers

SUMMARY:
This study evaluates the effect of different dietary conducts in the nocturnal period on the postprandial metabolism and food perceptions of night workers of the Hospital of Clinics of Uberlândia, Federal University of Uberlândia.

DETAILED DESCRIPTION:
Due to imbalances in the circadian rhythm, shift workers may present inadequate eating habits, which provoke metabolic and nutritional disorders. In this crossover study the participants consumed, at different times and separated by 6 days interval, two meals pre-established at the time of night work: a control and a higher-protein. On the day of each intervention, the participants were evaluated for response of blood and subjective markers after meal (glucose, insulin, triglycerides and subjective perceptions related to ingestion after each meal). It is expected that the standardization of a glycemic reduction diet will improve the metabolic response of the workers, demonstrated in the results of the biochemical parameters. If this scenario is confirmed, it is still expected that the data and results obtained in this study may serve as subsidies for the elaboration of nutritional interventions consistent with the work routine at night.

ELIGIBILITY:
Inclusion Criteria:

* Male workers;
* Age between 20 and 60 years;
* Have been working night shift for at least six months;
* Sedentary.

Exclusion Criteria:

* Failure to provide the information or material necessary for the development of the study;
* Carriers of diseases previously diagnosed and under treatment, such as type 2 diabetes mellitus, hypertension, cardiovascular diseases and related mood disorders such as depression.

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2018-01-11 (Actual); Study Completion 2018-01-11 (Actual)

PRIMARY OUTCOMES:
Change of metabolic parameters | 7 months
  Blood samples were collected before and after (30, 60, 90 and 120 minutes) the consumption of each of the meals at nighttime (work schedule). In the first meal of the following day (standard breakfast) were determined the serum concentrations of glucose (mg/dL).
Change of metabolic parameters | 7 months
  Blood samples were collected before and after (30, 60, 90 and 120 minutes) the consumption of each of the meals at nighttime (work schedule). In the first meal of the following day (standard breakfast) were determined the serum concentrations of insulin (mU/mL).
Change of metabolic parameters | 7 months
  Blood samples were collected before and after (30, 60, 90 and 120 minutes) the consumption of each of the meals at nighttime (work schedule). In the first meal of the following day (standard breakfast) were determined the serum concentrations of triglycerides (mg/dL).
Change of food perceptions | 7 months
  To evaluate appetite, satiety and postprandial satisfaction, a visual analogue scale called "hunger and satiety scale" was applied before and after consumption of the proposed meal, with the questions, "How much hunger did you have before the meal?"; "After the meal, how did you feel?"; "How much did you like the meal?", signaling all responses on a 0 to 10 cm scale. There is no classification of the values obtained. The answers are subjective and used in a comparative way.

CONTACTS AND LOCATIONS:
Overall Officials: CIBELE A CRISPIM, PhD, Principal Investigator — Federal University of Uberlandia
Locations (1):
- Cibele Aparecida Crispim, Uberlândia, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cunha NB, Silva CM, Mota MC, Lima CA, Teixeira KRC, Cunha TM, Crispim CA. A High-Protein Meal during a Night Shift Does Not Improve Postprandial Metabolic Response the Following Breakfast: A Randomized Crossover Study with Night Workers. Nutrients. 2020 Jul 13;12(7):2071. doi: 10.3390/nu12072071. PMID 32668588